CLINICAL TRIAL: NCT01776125
Title: Genetic Evaluation for the Scoliosis Gene(s) in Patients With Neurofibromatosis 1 and Scoliosis
Brief Title: Genetic Evaluation of NF1 and Scoliosis Patients
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Children Hospital Cincinnati OH (Unknown); Texas Scottish Rite Hospital for Children (Other); Norton Leatherman Spine Center (Other); Mayo Clinic (Other); University of Utah (Other); Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: 0804M30543
Record Dates: First submitted 2012-11-13; First posted 2013-01-25 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Neurofibromatosis 1; Scoliosis
Keywords: Neurofibromatosis Type One; Scoliosis
MeSH Terms: conditions — Neurofibromatosis 1; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Participants will be asked to give us a swab (a long Q-tip) of the inside of your cheek (inside your mouth) for genetic testing. This should take no more than 10 seconds. It will not hurt. The swab kit will be provided by Axial Biotech Inc. It will include a self-addressed stamped envelope to mail the swab back to Axial Biotech Inc. Participatns existing x-rays will be reviewed as part of this study as well. We will review participant's medical record to look at what treatments have been executed during the course of participation. Once the individual agrees to participate in this project their private health information will be sent to Axial Biotech Inc., the company that will be doing the genetic testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dystrophic Scolisis and NF1: Patients with NF1 diagnosed with dystrophic scoliosis that have been clinically treated will be asked for a cheek swab for genetic testing
  Interventions: Other: Cheek swab
- Non-dystrophic scoliosis and NF1: NF1 patients with non-dystrophic scoliosis that have been treated clinically. will be asked for a cheek swab for genetic testing
  Interventions: Other: Cheek swab

INTERVENTIONS:
Other: Cheek swab — Participants will be asked to give us a swab (a long Q-tip) of the inside of your cheek (inside your mouth) for genetic testing. This should take no more than 10 seconds. It will not hurt. The swab kit will be provided by Affiliated Genetics. It will include a self-addressed stamped envelope to mail the swab back to Affiliated Genetics. Participants existing x-rays will be reviewed as part of this study as well. We will review participant's medical record to look at what treatments have been executed during the course of participation. Once the individual agrees to participate in this project their private health information will be sent to Axial Biotech Inc., the company that will be doing the genetic testing.

SUMMARY:
Neurofibromatosis (NF) is a common genetic disorder that cause tumors to grow along various types of nerves and, in addition, can affect the development of bones and skin. It occurs in 1:4000 persons. NF has been classified into three distinct types: NF1, NF2 and Schwannomatosis. NF1 is the focus of this study.

NF1 is an extremely variable disorder which ranges from extremely mild cases in which the only signs of the disorder in adulthood may be multiple café-au-lait spots and a few dermal neurofibromas, to more severe cases like disfigurement, scoliosis and learning disabilities. Scoliosis (abnormal curvature of the spine) is perhaps the most common bone deformity in NF1 which usually appears in early childhood. There are two types: dystrophic and non-dystrophic scoliosis. Dystrophic scoliosis is usually associated with other bone deformities which are seen on x-ray and carries a poorer prognosis than non dystrophic scoliosis. There is evidence that genes other than the NF1 gene are responsible for the variable severity of cases. Recent studies have identified genetic markers for another condition called adolescent idiopathic scoliosis (scoliosis which presents in adolescent age group with no known cause). We believe that the same genetic markers may also be present in NF1 patients with scoliosis.

Our objective is primarily to determine if the same genetic markers discovered in adolescent idiopathic scoliosis are also present in NF1 patients with scoliosis.

DETAILED DESCRIPTION:
NF 1 patients with scoliosis can present as either non dystrophic or dystrophic scoliosis. Non dystrophic scoliosis behaves and evolves similarly to that of AIS patients. Therefore, we hypothesize that Neurofibromatosis type 1 patients with non-dystrophic scoliosis have a similar curve progression risk profile markers as patients with Adolescent Idiopathic Scoliosis. Dystrophic scoliosis patients will not have the same curve progression risk profile as AIS. The long range goal of this study is to possibly develop a genetic test in NF1 patients with scoliosis that is predictive of dystrophic or non-dystrophic type. The short term goal for the study is to see if the non-dystrophic curves have the same single-nucleotide polymorphisms (SNPs') as in AIS and if these SNPs are prognostic.

One of the goals of this study is to develop and validate a grading scheme to classify dystrophic changes in patients with NF 1 scoliosis. Radiographic characteristics of dystrophic deformity described by Crawford and Durrani et. al. will distinguish dystrophic scoliosis from non-dystrophic scoliosis. In addition, we will be performing genetic testing on patients with NF 1 who have had clinical treatment for scoliosis. Although the NF1 gene has been identified no specific genetic markers have been identified in NF1 patients with scoliosis. Genetic evaluation on a known group of NF1 patients with scoliosis will allow us to gain insight as to which phenotypes of NF1 patients would possibly develop spine deformities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Neurofibromatosis type 1 (NIH criteria)[24]
* Proper preoperative radiographs of the spine
* Spinal fusion done for scoliosis
* Age 8 to 65 years old

Exclusion Criteria:

* Paraspinal tumors causing scoliosis
* Patients who are unavailable to donate a swab sample for genetic testing will be excluded.

Enrollment Criteria:

* In general participants of this study should be NF1 patients with scoliosis who have either reached skeletal maturity or required surgical treatment.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Candidates will be identified by spine surgeons who are members of the Spinal Deformity Study Group. Participants need to be age 8 to 65 years old. These will be individuals who have been clinically diagnosed with NF 1 and have undergone spinal fusion for scoliosis (either dystrophic or non-dystrophic). The participating physicians will explain the research to qualifying patients or their guardians. We have added a flyer for the participating physicians to hand out to their patients. The patient/guardian may then take this flyer home and contact study personnel directly, thus removing the participating physician and/or his staff from the process.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
SCOLISCORE | 1 month after sample submission
  The SCOLISCORE Test is the first and only genetic test proven to give physicians and parents insight into the possible progression of patient with Adolescent Idiopathic Scoliosis (AIS), thereby reducing the uncertainty of AIS progression.

CONTACTS AND LOCATIONS:
Overall Officials: David W Polly, MD, Principal Investigator — University of Minnesota, Orthopaedic Surgery
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No